CLINICAL TRIAL: NCT01280591
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Trial Assessing the Efficacy of Naproxen Sodium and Diphenhydramine Combination in Postsurgical Dental Pain With Phase Advanced Sleep
Brief Title: Evaluate Analgesic/Sedative Efficacy of Naproxen Sodium and Diphenhydramine in Patients With Postsurgical Dental Pain
Acronym: Morpheus II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14837
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Pain, Postoperative
Keywords: Naproxen sodium; Diphenhydramine
MeSH Terms: conditions — Pain, Postoperative | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Naproxen sodium 440 mg / DPH 50 mg (BAY98-7111) (Experimental)
  Interventions: Drug: Naproxen sodium 440 mg / DPH 50 mg (BAY98-7111)
- Naproxen sodium 220 mg / DPH 50 mg (BAY98-7111) (Experimental)
  Interventions: Drug: Naproxen sodium 220 mg / DPH 50 mg (BAY98-7111)
- Naproxen sodium 440 mg (BAYH6689) (Active Comparator)
  Interventions: Drug: Naproxen sodium 440 mg (BAYH6689)
- DPH 50 mg (Active Comparator)
  Interventions: Drug: DPH 50 mg

INTERVENTIONS:
Drug: Naproxen sodium 440 mg / DPH 50 mg (BAY98-7111) — Participants received two Naproxen sodium 220 mg / DPH (Diphenhydramine hydrochloride) 25 mg tablets orally, single dose
  Arms: Naproxen sodium 440 mg / DPH 50 mg (BAY98-7111)
Drug: Naproxen sodium 220 mg / DPH 50 mg (BAY98-7111) — Participants received one Naproxen sodium 220 mg / DPH 50 mg tablet and one matching placebo capsule orally, single dose
  Arms: Naproxen sodium 220 mg / DPH 50 mg (BAY98-7111)
Drug: Naproxen sodium 440 mg (BAYH6689) — Participants received two Naproxen sodium 220 mg tablets orally, single dose
  Arms: Naproxen sodium 440 mg (BAYH6689)
Drug: DPH 50 mg — Participants received two DPH (Diphenhydramine hydrochloride) 25mg tablets orally, single dose
  Arms: DPH 50 mg

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of a single oral dose of two dose combinations of naproxen sodium and diphenhydramine (DPH) to demonstrate that naproxen sodium/DPH combination provides added clinical benefit to sleep improvement than either single ingredient alone in subjects with post-surgical dental pain and phase advanced sleep.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers ages 12 and older
* Scheduled to undergo surgical removal of a minimum of two third molars of which at least one has to be a mandibular third molar. The mandibular extraction(s) required by each subject must meet one of the following scenarios:

  * one full bony impaction
  * two partial bony impactions
  * one full bony impaction and one partial bony impaction
  * one full bony impaction and one soft tissue impaction
  * one full bony impaction and one erupted third molar. Two full bony mandibular impactions are not allowed. Maxillary third molars may be removed regardless of impaction level.
* Have moderate to severe postoperative pain on the Categorical Pain Rating Scale and a score of ≥ 50 mm on the 100-mm visual analog Pain Severity Rating Scale between 1600 hour and 1830 hour on the day of surgery
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, Depo-Provera, or double-barrier and have a negative pregnancy test at Screening and prior to surgery. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial, (subjects <18 years of age must sign a written assent and have parental or guardian consent).

Exclusion Criteria:

* History of hypersensitivity to naproxen, diphenhydramine, nonsteroidal anti-inflammatory drug (NSAIDS), tramadol, aspirin or any other antihistamine and similar pharmacological agents or components of the products
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than 50 percent obstruction (polyposis nasi, marked septal deviation) that can interfere with the conduct of the study in the judgment of the investigator
* Current or past history of bleeding disorder(s)
* Acute illness or local infection prior to surgery that can interfere with the conduct of the study in the judgment of the investigator
* Chronic use of antihistamines defined as using 5 or more times a week for 2 or more consecutive weeks during the past 3 months
* Positive alcohol breathalyzer test and positive urine drug test prior to surgery
* Females who are pregnant or lactating
* Chronic or severe sleep problems that do not respond to / Over the Counter (OTC) medication and requires a prescription hypnotic or sedative
* Habitually spends less than 6.5 hours in bed

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 712 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Austin, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Cooper S, Laurora I, Wang Y, Venkataraman P, An R, Roth T. Efficacy and tolerability studies evaluating a sleep aid and analgesic combination of naproxen sodium and diphenhydramine in the dental impaction pain model in subjects with induced transient insomnia. Int J Clin Pract. 2015 Oct;69(10):1149-58. doi: 10.1111/ijcp.12669. Epub 2015 May 21. PMID 25996289

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Started | 203 | 204 | 203 | 102
Completed | 203 | 204 | 203 | 99
Not Completed | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Does not meet exclusion #27 criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg | Total
Number analyzed (Participants) | 203 | 204 | 203 | 102 | 712
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.4 (4.87) | 21.0 (4.25) | 21.0 (4.50) | 21.5 (5.59) | 21.2 (4.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 124 | 117 | 54 | 403
  Male | 95 | 80 | 86 | 48 | 309
Baseline Categorical Pain Rating Scale [Number; unit: Participants]
  No pain | 0 | 0 | 0 | 0 | 0
  Mild pain | 0 | 0 | 0 | 0 | 0
  Moderate pain | 146 | 134 | 140 | 74 | 494
  Severe pain | 57 | 70 | 63 | 28 | 218

OUTCOME MEASURES:

1. Primary Outcome: Wake Time After Sleep Onset (WASO) Measured by Actigraphy
Description: WASO was defined as Total wake time (in minutes) after sleep onset during the 10 hours in-bed period as measured by actigraphy. Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 203 | 102
Minutes | 143.7 [117.9 to 169.6] | 230.9 [205.2 to 256.5] | 214.0 [188.2 to 239.8] | 431.4 [395.1 to 467.6]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -70.3, 95% CI 2-sided [-106.8 to -33.7], Standard Error of Mean 13.17

2. Primary Outcome: Sleep Latency Measured by Actigraphy
Description: Sleep latency was defined as the time to sleep onset from the time of dosing as measured by actigraphy. Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 203 | 102
Minutes | 25.50 [22.50 to 30.00] | 30.25 [25.00 to 33.50] | 25.75 [22.50 to 29.50] | 41.50 [26.50 to 54.50]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs DPH 50 mg; Test type: Superiority or Other; p < 0.0001, Log Rank

3. Secondary Outcome: Total Sleep Time Measured by Actigraphy
Description: Total time time was measured as total time spent sleeping (not to exceed 600 minutes) during the in-bed period as measured by actigraphy. Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 203 | 102
Minutes | 426.2 [400.9 to 451.4] | 337.7 [312.6 to 362.7] | 355.8 [330.6 to 381.0] | 141.4 [106.0 to 176.8]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = 70.4, 95% CI 2-sided [28.1 to 112.7], Standard Error of Mean 12.85

4. Secondary Outcome: Sleep Efficiency Measured by Actigraphy
Description: Sleep efficiency was calculated as (total sleep time/total time in-bed time) × 100; total in-bed time was fixed at 10 hours. Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of sleep time during in-bed time
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 203 | 102
Percent of sleep time during in-bed time | 71.0 [66.8 to 75.2] | 56.3 [52.1 to 60.5] | 59.3 [55.1 to 63.5] | 23.6 [17.7 to 29.5]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = 11.7, 95% CI 2-sided [3.7 to 19.7], Standard Error of Mean 2.14

5. Secondary Outcome: Global Assessment of Investigational Product as a Sleep Aid
Description: The Global Assessment of Investigational Product as a Sleep-Aid was rated using a 5-point categorical scale for which the potential response was poor (0), fair, (1), good (2), very good (3), or excellent (4).
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 166 | 125 | 141 | 25
Participants
  0 = Poor | 8 | 10 | 29 | 3
  1 = Fair | 39 | 29 | 51 | 9
  2 = Good | 58 | 47 | 37 | 6
  3 = Very good | 49 | 26 | 17 | 7
  4 = Excellent | 12 | 13 | 7 | 0
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Karolinska Sleep Diary - Sleep Quality
Description: Subjects responded to the following question: How was your sleep? very poor (1); rather poor (2); neither poor nor good (3); rather good (4); very good (5)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Participants
  1 = Very poor | 3 | 5 | 5 | 3
  2 = Rather poor | 23 | 24 | 39 | 10
  3 = Neither poor nor good | 46 | 52 | 69 | 13
  4 = Rather good | 82 | 68 | 55 | 18
  5 = Very good | 34 | 21 | 12 | 2
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0027, Cochran-Mantel-Haenszel

7. Secondary Outcome: Karolinska Sleep Diary - Calmness of Sleep
Description: Subjects responded to the following question: How calm was your sleep? very restless (1); rather restless (2); neither restless nor calm (3); rather calm (4); very calm (5)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Participants
  1 = Very restless | 8 | 8 | 7 | 5
  2 = Rather restless | 35 | 29 | 48 | 16
  3 = Neither restless nor calm | 37 | 39 | 42 | 10
  4 = Rather calm | 76 | 68 | 61 | 12
  5 = Very calm | 32 | 26 | 22 | 3
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0321, Cochran-Mantel-Haenszel

8. Secondary Outcome: Karolinska Sleep Diary - Easiness to Fall Asleep
Description: Subjects responded to the following question: How easy was it to fall asleep? very difficult (1); rather difficult (2); neither difficult nor easy (3); rather easy (4); very easy (5)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Participants
  1 = Very difficult | 8 | 11 | 12 | 8
  2 = Rather difficult | 41 | 45 | 59 | 16
  3 = Neither difficult nor easy | 57 | 57 | 55 | 10
  4 = Rather easy | 62 | 42 | 41 | 9
  5 = Very easy | 20 | 15 | 13 | 3
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel

9. Secondary Outcome: Karolinska Sleep Diary - Premature Awakening
Description: Subjects responded to the following question: Premature awakening? woke up much too early (1); woke up somewhat too early (2); no (3)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Participants
  1 = Woke up much too early | 40 | 54 | 65 | 23
  2 = Woke up somewhat too early | 77 | 59 | 80 | 17
  3 = No | 71 | 57 | 35 | 6
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

10. Secondary Outcome: Karolinska Sleep Diary - Ease of Awakening
Description: Subjects responded to the following question: Ease of awakening? (1) very difficult; (2) rather difficult; (3) neither difficult nor easy; (4) rather easy; very easy (5)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Participants
  1 = Very difficult | 0 | 0 | 1 | 0
  2 = Rather difficult | 7 | 4 | 2 | 1
  3 = Neither difficult nor easy | 28 | 24 | 33 | 10
  4 = Rather easy | 98 | 94 | 88 | 15
  5 = Very easy | 55 | 48 | 56 | 20
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p > 0.05, Cochran-Mantel-Haenszel

11. Secondary Outcome: Karolinska Sleep Diary - Well Rested
Description: Subjects responded to the following question: Well Rested? not rested at all (1); somewhat unrested (2); completely rested (3)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Participants
  1 = Not rested at all | 9 | 21 | 16 | 8
  2 = Somewhat unrested | 100 | 95 | 116 | 31
  3 = Completely rested | 79 | 54 | 48 | 7
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel

12. Secondary Outcome: Karolinska Sleep Diary - Sufficient Sleep
Description: Subjects responded to the following question: Did you get enough (sufficient) sleep? no, definitely too little (1); no, much too little (2); no, somewhat too little (3); yes, almost enough (4); yes, definitely enough (5)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Participants
  1 = No, definitely too little | 7 | 21 | 18 | 10
  2 = No, much too little | 14 | 24 | 22 | 8
  3 = No, somewhat too little | 37 | 40 | 56 | 14
  4 = Yes, almost enough | 84 | 52 | 58 | 9
  5 = Yes, definitely enough | 46 | 33 | 26 | 5
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

13. Secondary Outcome: Subjective Sleep Questionnaire - Quality of Your Sleep Last Night
Description: Subjects responded to Quality of sleep (10-point scale, where 1 was poor and 10 was excellent)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 183 | 162 | 174 | 45
Scores on a scale | 6.4 (1.96) | 5.9 (2.13) | 5.4 (1.99) | 4.9 (2.36)
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

14. Secondary Outcome: Subjective Sleep Questionnaire - Refreshing Nature of Your Sleep Last Night
Description: Subjects responded to Refreshing nature of sleep (10-point scale, where 1 was not refreshing and 10 was very refreshing)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 171 | 161 | 170 | 45
Scores on a scale | 6.2 (2.03) | 5.8 (2.26) | 5.5 (2.14) | 4.4 (2.45)
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0016, Cochran-Mantel-Haenszel

15. Secondary Outcome: Subjective Sleep Questionnaire - Time to Fall Asleep Last Night
Description: Subjects responded to Estimate of how long it took to fall asleep (minutes)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Minutes | 40.0 (31.52) | 40.7 (29.39) | 53.4 (67.78) | 42.4 (42.02)
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p > 0.05, Cochran-Mantel-Haenszel

16. Secondary Outcome: Subjective Sleep Questionnaire - Number of Minutes You Think That You Were Awake From the Time You Fell Asleep Until the Time You Got Out of Bed
Description: Subjects responded to Estimate of the amount of time the subject was awake from the time he or she fell asleep until the time he or she got out of bed (hours and minutes)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 188 | 170 | 180 | 46
Minutes | 73.8 (79.06) | 75.3 (81.55) | 103.5 (89.50) | 81.7 (86.72)
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

17. Secondary Outcome: Change From Baseline in Pain Intensity
Description: Pain Severity was collected on a 4-point categorical scale: 0=no pain, 1=mild pain, 2=moderate pain, 4=severe pain
Time Frame: Baseline and up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 203 | 102
Scores on a scale | -1.2 (1.01) | -0.7 (1.05) | -0.9 (0.99) | 0.1 (0.82)
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0064, ANCOVA

18. Secondary Outcome: Overall Rating of Pain Relief
Description: The Pain Relief Rating Scale was a 5-point categorical scale which included the following possible responses to the request to finish statement "Overall, the relief from my starting pain was": no relief (0); a little relief (1); some relief (2); a lot of relief (3); complete relief (4).
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 202 | 102
Participants
  0 = No relief | 44 | 89 | 68 | 79
  1 = A little relief | 4 | 4 | 8 | 1
  2 = Some relief | 32 | 29 | 24 | 11
  3 = A lot of relief | 65 | 53 | 62 | 8
  4 = Complete relief | 58 | 29 | 40 | 3
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0047, Cochran-Mantel-Haenszel

19. Secondary Outcome: Time to Rescue Medication
Description: If rescue medication was taken by a subject for pain, then the time of rescue medication administration was recorded
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 203 | 102
Minutes | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | 113.5 [98.50 to 144.50]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.0053, Log Rank

20. Secondary Outcome: Cumulative Proportion of Subjects Taking Rescue Medication by Hour
Description: If rescue medication was taken by a subject for pain, then the time of rescue medication administration was recorded
Time Frame: Up to 10 hours
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 203 | 204 | 203 | 102
participants
  ≤ 60 minutes | 0 | 1 | 0 | 0
  ≤ 120 minutes | 18 | 36 | 27 | 53
  ≤ 180 minutes | 23 | 50 | 41 | 66
  ≤ 240 minutes | 25 | 57 | 47 | 70
  ≤ 300 minutes | 29 | 65 | 50 | 74
  ≤ 360 minutes | 34 | 69 | 55 | 76
  ≤ 420 minutes | 36 | 78 | 62 | 77
  ≤ 480 minutes | 39 | 83 | 63 | 78
  ≤ 540 minutes | 42 | 87 | 67 | 78
  ≤ 600 minutes | 43 | 89 | 68 | 78

21. Secondary Outcome: Global Assessment of Investigational Product as a Pain Reliever
Description: The Global Assessment of Investigational Product as a Pain Reliever was a 5- point categorical scale which included the following possible responses: poor (0); fair (1); good (2); very good (3); excellent (4).
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Number analyzed (Participants) | 166 | 126 | 141 | 25
Participants
  0 = Poor | 2 | 2 | 0 | 4
  1 = Fair | 9 | 16 | 15 | 5
  2 = Good | 43 | 35 | 36 | 9
  3 = Very good | 64 | 48 | 56 | 7
  4 = Excellent | 48 | 25 | 34 | 0
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.2734, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from the date of the first dose of study drug in the treatment period for 2 days, or for 30 days after the last study drug administration if they were serious adverse events (SAEs).
Arm/Group | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) | Naproxen Sodium 440 mg (BAYH6689) | DPH 50 mg
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/204 | 0/203 | 0/102
Other Adverse Events (participants affected / at risk) | 37/203 | 37/204 | 40/203 | 25/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naproxen Sodium 440 mg / DPH 50 mg (BAY98-7111) (N=203) | Naproxen Sodium 220 mg / DPH 50 mg (BAY98-7111) (N=204) | Naproxen Sodium 440 mg (BAYH6689) (N=203) | DPH 50 mg (N=102)
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 15 | 12 | 14 | 9
Vomiting (Gastrointestinal disorders) | 2 | 5 | 6 | 4
Chills (General disorders) | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 1 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 9 | 7 | 5 | 4
Headache (Nervous system disorders) | 12 | 13 | 15 | 8
Paraesthesia (Nervous system disorders) | 3 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 3 | 3 | 2 | 1
Syncope (Nervous system disorders) | 2 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No